CLINICAL TRIAL: NCT02438800
Title: Video Counseling for Effective Postpartum Contraception: a Randomized Clinical Trial
Brief Title: Video Counseling for Effective Postpartum Contraception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15-0665
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Contraception
Keywords: Postpartum Period

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Counseling (No Intervention): Women in this arm will receive standard contraceptive counseling routinely provided during prenatal care. All participants will receive information regarding access to free LARC methods in the postpartum period.
- Video Counseling (Experimental): Women in this arm will receive LARC First video-based contraceptive counseling in addition to standard contraceptive counseling routinely provided during prenatal care. All participants will receive information regarding access to free LARC methods in the postpartum period.
  Interventions: Behavioral: LARC First Video

INTERVENTIONS:
Behavioral: LARC First Video — LARC First is an evidence-based, 12-minute video developed by the CHOICE project that features women of all racial and ethnic backgrounds describing LARC methods of contraception in simple, understandable language with summary text when appropriate.
  Arms: Video Counseling

SUMMARY:
This is a randomized clinical trial to evaluate if the addition of long-acting reversible contraception (LARC) focused video-counseling during prenatal care increases uptake of postpartum LARC.

DETAILED DESCRIPTION:
Eligible participants will be identified in the prenatal period and will be randomized to one of two groups. The control group will receive the standard of care contraceptive counseling during prenatal counseling. The intervention group will also receive the standard of care contraceptive counseling during prenatal care, but will also watch an evidence-based,12 minute LARC First video created by the CHOICE project which provides information on different contraceptive methods. All participants will receive information regarding access to free LARC methods in the postpartum period. All participants will be called at 12 weeks postpartum. Independent of randomization arm, they will all undergo a 5-minute survey by phone about contraceptive method choice and use.

ELIGIBILITY:
Inclusion Criteria:

* woman presenting for routine prenatal care visit at University of North Carolina (UNC) Resident Continuity Clinic
* least 18 years old
* fluent in English
* able to read to a third-grade reading level
* not planning sterilization for postpartum contraception
* at least 28 weeks gestation at time of enrollment

Exclusion Criteria:

* those who do not meet the previously outlined inclusion criteria
* those who are unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of women who received an intrauterine device (IUD) or implant by 12 weeks postpartum | 12 weeks postpartum

SECONDARY OUTCOMES:
Proportion of women using any contraceptive method at 12 weeks postpartum | 12 weeks postpartum
Proportion of women who attended a postpartum visit | 12 weeks postpartum
Proportion of women answering agree or strongly agree to the following statement "I would recommend birth control counseling by video to a friend." | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Morse, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Women's Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided